CLINICAL TRIAL: NCT01201928
Title: A Phase 3b, Multicenter, Clinical Trial to Evaluate Pulmonary Function in a Subset of Subjects With Type 1 or Type 2 Diabetes
Brief Title: Pulmonary Function Substudy for Subjects Enrolled in Studies MKC-TI-161, MKC-TI-162 or MKC-TI-166
Status: Terminated | Type: Observational
Why Stopped: Parent trials were either not initiated or terminated
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MKC-TI-164
Record Dates: First submitted 2010-08-27; First posted 2010-09-15 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Technosphere Insulin Inhalation Powder
  Interventions: Drug: Technosphere Insulin Inhalation Powder
- Comparator: Based on parent trial
  Interventions: Drug: Comparator administered in parent trial

INTERVENTIONS:
Drug: Comparator administered in parent trial — Comparator arm may be different for each parent trial, consisting of some sort of usual care for diabetes
  Groups: Comparator
Drug: Technosphere Insulin Inhalation Powder — Pulmonary delivered inhaled insulin formulation containing human insulin and Technosphere Inhalation Powder (administered in parent trial)
  Groups: Technosphere Insulin Inhalation Powder

SUMMARY:
The purpose of this study is to evaluate pulmonary function test (PFT) sub-study in interested subjects from studies MKC-TI-161, MKC-TI-162 and MKC-TI-166. 100 Type I and 100 Type II diabetics will be enrolled. Each subject will undergo 6 PFT assessments over the course of the parent study.

DETAILED DESCRIPTION:
This study is designed to evaluate and compare changes in pulmonary function (FEV1(forced expiratory volume in 1 second) FVC(forced vital capacity), TLC (total lung capacity) and DLco) in subjects enrolled in 1 of 3 parent trials (MKC-TI-161, MKC-TI-162 or MKC-TI-166). Up to 100 subjects with Type I and Type II diabetes in the TI Inhalation Powder arm, and 100 subjects with Type I and Type II diabetes in the comparator arm will be enrolled. Each subject will undergo 6 PFT assessments over the course of the parent trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in one of three parent trials (MKC-TI-161, MKC-TI-162 or MKC-TI-166)

Exclusion Criteria:

* Subjects who are unable to perform PFTs that meet American Thoracic Society/European Respiratory Society (ATS/ERS) quality recommendations for acceptability and repeatability will be excluded from this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interested subjects enrolled in one of three parent trials; MKC-TI-161, MKC-TI-162 or MKC-TI-166
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Comparison of change from baseline to final treatment visit in pulmonary function (FEV1 FVC, TLC and DLco) between treatment Groups (TI vs comparator arms) using ANCOVA models. | Baseline values are the average of Visit 1 (Week -7) and Visit 4 (Week 0).

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Valley Research, Fresno, California
  - Health Care Partners Medical Group, Long Beach, California
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - LaPorte County Institute for Clinical Research Inc., Michigan City, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Endocrine Research Physicians East PA, Greenville, North Carolina
  - Israel Hartman MD, Arlington, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - SAM Clinical Research Center, San Antonio, Texas